CLINICAL TRIAL: NCT02625259
Title: A Phase 1, Open-Label Study to Evaluate the Relative Bioavailability, Effect of Food, and Gastric pH Modification on the Pharmacokinetics of MLN1117 in Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability, Effect of Food, and Gastric Potential Hydrogen (pH) Modification on the Pharmacokinetics of TAK-117 (MLN1117) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MLN1117-1002; U1111-1159-5909 (Registry Identifier: WHO)
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-07

CONDITIONS: Neoplasm, Advanced or Metastatic
Keywords: Drug therapy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — serabelisib; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: TAK-117 9*100 mg + TAK-117 3*300 mg (Experimental): TAK-117900 milligram (mg), capsules, orally, once on Day 1, followed by 2 weeks of washout, followed by TAK-117 900 mg, tablets, orally, once on Day 15.
  Interventions: Drug: TAK-117
- Part 1: TAK-117 3*300 mg + TAK-117 9*100 mg (Experimental): TAK-117 900 mg tablets, orally, once on Day 1, followed by 2 weeks of washout, followed by TAK-117 900 mg, capsules, orally, once on Day 15.
  Interventions: Drug: TAK-117
- Part 2: TAK-117 Fasted + TAK-117 Fed (Experimental): TAK-117 at the dose determined in Part 1, tablets, in fasted condition, orally, once on Day 1, followed by 2 weeks of washout, followed by TAK-117 at the dose determined in Part 1, tablets, with a standard high-fat meal, orally, once on Day 15.
  Interventions: Drug: TAK-117
- Part 2: TAK-117 Fed + TAK-117 Fasted (Experimental): TAK-117 at the dose determined in Part 1, tablets, with a standard high-fat meal, orally, once on Day 1, followed by 2 weeks of washout, followed by TAK-117 at the dose determined in Part 1, tablets, in fasted condition, orally, once on Day 15.
  Interventions: Drug: TAK-117
- Part 3: TAK-117 + Lansoprazole (Experimental): TAK-117 at the dose determined in Part 1, tablets, orally, once on Day 1, followed by lansoprazole 30 mg, tablets or capsules, once daily from Day 10 to Day 15, followed by TAK-117 at the dose determined in Part 1, tablets, orally, once on Day 15.
  Interventions: Drug: Lansoprazole; Drug: TAK-117

INTERVENTIONS:
Drug: TAK-117 — TAK-117 capsules
  Arms: Part 1: TAK-117 3*300 mg + TAK-117 9*100 mg; Part 1: TAK-117 9*100 mg + TAK-117 3*300 mg
Drug: Lansoprazole — Lansoprazole capsules
  Arms: Part 3: TAK-117 + Lansoprazole
Drug: TAK-117 — TAK-117 tablets

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of a new tablet formulation of TAK-117 (new clinical trial material [NTM]) compared to the TAK-117 Process B capsules (current clinical trial material [CTM]) (Part 1), to assess the effects of food on the oral bioavailability and pharmacokinetics (PK) of TAK-117 (Part 2), and to assess the effects of gastric pH-modifying agent on the PK of TAK-117 in healthy participants (Part 3).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-117. TAK-117 is being tested to treat people who have advanced solid tumors. This study will look at the PK and relative bioavailability of new tablet formulation of TAK-117 as compare to current capsule formulation in Part 1. In Part 2 and Part 3, interaction of TAK-117 with food and a gastric pH modifying agent will be evaluated respectively in healthy participants, and will commence only after the completion of Part 1.

The study will enroll approximately 54 participants. In Part 1, participants will be randomly assigned (by chance, like flipping a coin) to 1 of the 2 crossover sequences:

* Sequence A: TAK-117 capsules (9*100 mg) first then TAK-117 tablets (3*300 mg)
* Sequence B: TAK-117 tablets (3*300 mg) first then TAK-117 capsules (9*100 mg)

Part 2 and Part 3 will be evaluated only on the new tablet formulation of TAK-117 at the dose determined in Part 1. In Part 2, participants will be randomly assigned to receive a single dose of TAK-117 in the fasted state followed by TAK-117 with standard high-fat breakfast in Sequence A or vice-versa in Sequence B. In Part 3, participants will receive a single dose of TAK-117 on Day 1 followed by lansoprazole 30 mg on Day 10 for 6 days and then second dose of TAK-117 on Day 15. Blood samples will be collected at predose and up to 72 hours postdose at prespecified time points on Days 1 and 15. Urine samples will be collected predose, 0 to 12 hours, and 12 to 24 hours postdose in Part 1 only.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 45 days. Participants will make 2 visits to the clinic in each part, during which they will remain confined to the clinic for a 4 to 10 day period for drug dosing and other study procedures. Participants will also complete a final visit 30 to 33 days after their last dose of study drug for a follow-up assessment (Day 45).

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 18 to 45 years inclusive, at the time of consent.
2. Is healthy adult male or female.
3. Weighs greater than or equal to (>=) 45 kilogram (kg) (female) or >=55 kg (male), and body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive, at screening.
4. Suitable venous access for the study-required blood sampling, including PK sampling.
5. Has provided the voluntary written consent.

Exclusion Criteria:

1. Any clinically significant abnormality at screening or medical history of cardiac, hepatic, renal, respiratory, gastrointestinal (GI), endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
2. Manifestations of malabsorption due to prior GI surgery, GI disease, or for an unknown other reason that may alter the PK of TAK-117 or lansoprazole.
3. Creatinine clearance less than or equal to (<=) 90 milliliter per minute (mL/min) based either on Cockroft-Gault estimate or based on a 12- or 24-hour urine collection during screening.
4. Known intolerance to TAK-117 or lansoprazole, or any of the excipients of either drug.
5. A positive test result for human immunodeficiency virus (HIV), hepatitis A antibody (HAVAb), hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibody Anti-HBc (IgM), or hepatitis C antibody (HCVAb) tests at screening, or serological reactions for syphilis during screening.
6. Has Lactose intolerance (only for Part 2).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2016-05-16 (Actual); Study Completion 2016-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 08 January 2016 to 22 July 2016.
Pre-assignment Details: Healthy participants were enrolled in this 3-part study to receive TAK-117 in Part 1 as: Crossover of 9*100 milligram (mg) capsules or 3*300 mg tablets, Part 2: Crossover of TAK-117 in fasted or fed state and Part 3: TAK-117 with lansoprazole.
Groups:
- Part-1: TAK-117 900 mg Capsules + TAK-117 900 mg Tablets: TAK-117 9*100 mg, capsules (current clinical trial material [CTM]), orally, once on Day 1 (first intervention), followed by washout from Day 2 to Day 14, further followed by TAK-117 3*300 mg, tablets (new clinical trial material [NTM]), orally, once on Day 15 (second intervention).
- Part-1: TAK-117 900 mg Tablets + TAK-117 900 mg Capsules: TAK-117 3*300 mg, tablets (NTM), orally, once on Day 1 (first intervention), followed by washout from Day 2 to Day 14, further followed by TAK-117 9*100 mg, capsules (CTM), orally, once on Day 15 (second intervention).
- Part-2: TAK-117 600 mg Fasted + TAK-117 600 mg Fed: TAK-117 2*300 mg, tablets (NTM), orally, once in the fasted state on Day 1 (first intervention), followed by washout from Day 2 to Day 14, further followed by TAK-117 2*300 mg, tablets (NTM), orally, with a standard high-fat breakfast, once on Day 15 (second intervention).
- Part-2: TAK-117 600 mg Fed + TAK-117 600 mg Fasted: TAK-117 2*300 mg, tablets (NTM), orally, once with a standard high-fat breakfast on Day 1 (first intervention), followed by washout from Day 2 to Day 14, further followed by TAK-117 2*300 mg, tablets (NTM), orally, in the fasted state, once on Day 15 (second intervention).
- Part-3: TAK-117 900 mg + Lansoprazole 30 mg: TAK-117 3*300 mg, tablets (NTM), orally, once on Day 1, followed by lansoprazole 30 mg, capsule, orally, once daily from Day 10 to Day 15 along with TAK-117 3*300 mg, tablets (NTM), orally, once on Day 15 approximately 1 hour (hr) after the last dose of lansoprazole 30 mg.
Period: First Intervention (Day 1)
Arm/Group | Part-1: TAK-117 900 mg Capsules + TAK-117 900 mg Tablets | Part-1: TAK-117 900 mg Tablets + TAK-117 900 mg Capsules | Part-2: TAK-117 600 mg Fasted + TAK-117 600 mg Fed | Part-2: TAK-117 600 mg Fed + TAK-117 600 mg Fasted | Part-3: TAK-117 900 mg + Lansoprazole 30 mg
Started | 11 | 9 | 8 | 10 | 16
Completed | 9 | 8 | 7 | 9 | 16
Not Completed | 2 | 1 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Washout (Day 2 to Day 14)
Arm/Group | Part-1: TAK-117 900 mg Capsules + TAK-117 900 mg Tablets | Part-1: TAK-117 900 mg Tablets + TAK-117 900 mg Capsules | Part-2: TAK-117 600 mg Fasted + TAK-117 600 mg Fed | Part-2: TAK-117 600 mg Fed + TAK-117 600 mg Fasted | Part-3: TAK-117 900 mg + Lansoprazole 30 mg
Started | 9 | 8 | 7 | 9 | 0
Completed | 9 | 8 | 7 | 9 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Day 15)
Arm/Group | Part-1: TAK-117 900 mg Capsules + TAK-117 900 mg Tablets | Part-1: TAK-117 900 mg Tablets + TAK-117 900 mg Capsules | Part-2: TAK-117 600 mg Fasted + TAK-117 600 mg Fed | Part-2: TAK-117 600 mg Fed + TAK-117 600 mg Fasted | Part-3: TAK-117 900 mg + Lansoprazole 30 mg
Started | 9 | 8 | 7 | 9 | 0
Completed | 9 | 8 | 7 | 9 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all the participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part-1: TAK-117 900 mg Capsules + TAK-117 900 mg Tablets | Part-1: TAK-117 900 mg Tablets + TAK-117 900 mg Capsules | Part-2: TAK-117 600 mg Fasted + TAK-117 600 mg Fed | Part-2: TAK-117 600 mg Fed + TAK-117 600 mg Fasted | Part-3: TAK-117 900 mg + Lansoprazole 30 mg | Total
Number analyzed (Participants) | 11 | 9 | 8 | 10 | 16 | 54
Age, Customized [Number; unit: participants]
  18-45 years | 11 (7.63) | 9 (7.79) | 8 (7.15) | 10 (6.13) | 16 (6.88) | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 4 | 10 | 9 | 38
  Male | 3 | 2 | 4 | 0 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 4 | 4 | 6 | 24
  Not Hispanic or Latino | 5 | 5 | 4 | 6 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 3 | 8 | 19
  White | 8 | 5 | 4 | 7 | 5 | 29
  More than one race | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 8 | 10 | 16 | 54

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-117
Time Frame: Part 1 and 2: Day 1 or 15 pre-dose and at multiple time points (up to 72 hours) post-dose; Part 3: Day 1 (TAK-117) and Day 15 (TAK-117 + Lansoprazole) pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK)-evaluable population included participants who received both doses of TAK-117 study drug in each sequence and had sufficient PK data to reliably estimate PK parameters that were used for PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules): TAK-117 9*100 mg, capsules (CTM), orally, once on Day 1 or 15 of intervention period.
- Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets): TAK-117 3*300 mg, tablets (NTM), orally, once on Day 1 or 15 of intervention period.
- Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets): TAK-117 2*300 mg, tablets (NTM), orally, once in a fasted state on Day 1 or 15 of intervention period.
- Part-2: TAK-117 600 mg Fed (2*300 mg Tablets): TAK-117 2*300 mg, tablets (NTM), orally, with a standard high-fat breakfast, once on Day 1 or 15 of intervention period.
- Part-3: TAK-117 900 mg (3*300 mg Tablets): TAK-117 3*300 mg, tablets (NTM), orally, once on Day 1.
- Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg: Lansoprazole 30 mg, capsule, orally, once daily from Day 10 to Day 15 along with TAK-117 3*300 mg, tablets (NTM), orally once on Day 15.
Arm/Group | Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) | Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets) | Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) | Part-2: TAK-117 600 mg Fed (2*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg
Number analyzed (Participants) | 17 | 17 | 16 | 16 | 16 | 16
nanogram per milliliter (ng/mL) | 4632.992 (71) | 6225.347 (53) | 6455.111 (48) | 7847.591 (24) | 5859.156 (58) | 190.172 (144)
Statistical Analysis 1: Comparison: Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) vs Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets); Analysis of variance was performed for calculating 90 percent (%) confidence intervals (CIs) for the ratios of log-transformed geometric mean Cmax of TAK-117 tablet versus capsule dosage form; Test type: Superiority or Other; Geometric mean ratio = 1.36, 90% CI 2-sided [1.00 to 1.83]
Statistical Analysis 2: Comparison: Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) vs Part-2: TAK-117 600 mg Fed (2*300 mg Tablets); Analysis of variance was performed for calculating 90% CIs for the ratios of log-transformed geometric mean Cmax of TAK-117 tablet dosage form with food versus without food; Test type: Superiority or Other; Geometric mean ratio = 1.20, 90% CI 2-sided [0.86 to 1.67]
Statistical Analysis 3: Comparison: Part-3: TAK-117 900 mg (3*300 mg Tablets) vs Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg; Analysis of variance was performed for calculating 90% CIs for the ratios of log-transformed geometric mean Cmax of TAK-117 tablet dosage form with lansoprazole versus a single dose of TAK-117 alone; Test type: Superiority or Other; Geometric mean ratio = 0.03, 90% CI 2-sided [0.02 to 0.07]

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-117
Time Frame: as for outcome 1
Population: The PK-evaluable population included participants who received both doses of TAK-117 study drug in each sequence and had sufficient PK data to reliably estimate PK parameters that were used for PK analyses.
Measure: Median (Full Range); unit: hours
Arm/Group | Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) | Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets) | Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) | Part-2: TAK-117 600 mg Fed (2*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg
Number analyzed (Participants) | 17 | 17 | 16 | 16 | 16 | 16
hours | 2.067 [1.00 to 6.00] | 3.000 [0.500 to 6.00] | 3.000 [2.00 to 6.07] | 6.033 [4.00 to 8.03] | 3.000 [1.00 to 6.00] | 3.517 [1.00 to 6.00]

3. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-117
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) | Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets) | Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) | Part-2: TAK-117 600 mg Fed (2*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg
Number analyzed (Participants) | 17 | 17 | 16 | 16 | 16 | 16
nanogram*hour per milliliter (ng*hr/mL) | 45727.280 (94) | 66015.952 (91) | 71442.968 (67) | 127143.511 (39) | 63165.064 (91) | 1018.650 (129)
Statistical Analysis 1: Comparison: Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) vs Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets); Analysis of variance was performed for calculating 90 % CIs for the ratios of log-transformed geometric mean AUClast of TAK-117 tablet versus capsule dosage form; Test type: Superiority or Other; Geometric mean ratio = 1.47, 90% CI 2-sided [0.98 to 2.18]
Statistical Analysis 2: Comparison: Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) vs Part-2: TAK-117 600 mg Fed (2*300 mg Tablets); Analysis of variance was performed for calculating 90% CIs for the ratios of log-transformed geometric mean AUClast of TAK-117 tablet dosage form with food versus without food; Test type: Superiority or Other; Geometric mean ratio = 1.76, 90% CI 2-sided [1.11 to 2.78]
Statistical Analysis 3: Comparison: Part-3: TAK-117 900 mg (3*300 mg Tablets) vs Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg; Analysis of variance was performed for calculating 90% CIs for the ratios of log-transformed geometric mean AUClast of TAK-117 tablet dosage form with lansoprazole versus a single dose of TAK-117 alone; Test type: Superiority or Other; Geometric mean ratio = 0.02, 90% CI 2-sided [0.01 to 0.04]

4. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-117
Time Frame: as for outcome 1
Population: The PK-evaluable population where data at specified time points were available. The PK-evaluable population included participants who received both doses of TAK-117 study drug in each sequence and had sufficient PK data to reliably estimate PK parameters that were used for PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) | Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets) | Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) | Part-2: TAK-117 600 mg Fed (2*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) | Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg
Number analyzed (Participants) | 13 | 13 | 15 | 16 | 15 | 4
ng*hr/mL | 64165.340 (77) | 96293.083 (77) | 81595.634 (61) | 128336.896 (39) | 85782.122 (85) | 6547.254 (66)
Statistical Analysis 1: Comparison: Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) vs Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets); Analysis of variance was performed for calculating 90 % CIs for the ratios of log-transformed geometric mean AUC∞ of TAK-117 tablet versus capsule dosage form; Test type: Superiority or Other; Geometric mean ratio = 1.53, 90% CI 2-sided [0.93 to 2.51]
Statistical Analysis 2: Comparison: Part-2: TAK-117 600 mg Fasted (2*300 mg Tablets) vs Part-2: TAK-117 600 mg Fed (2*300 mg Tablets); Analysis of variance was performed for calculating 90% CIs for the ratios of log-transformed geometric mean AUC∞ of TAK-117 tablet dosage form with food versus without food; Test type: Superiority or Other; Geometric mean ratio = 1.50, 90% CI 2-sided [1.00 to 2.25]
Statistical Analysis 3: Comparison: Part-3: TAK-117 900 mg (3*300 mg Tablets) vs Part-3: TAK-117 900 mg (3*300 mg Tablets) + Lansoprazole 30 mg; Analysis of variance was performed for calculating 90% CIs for the ratios of log-transformed geometric mean AUC∞ of TAK-117 tablet dosage form with lansoprazole versus a single dose of TAK-117 alone; Test type: Superiority or Other; Geometric mean ratio = 0.08, 90% CI 2-sided [0.03 to 0.18]

5. Secondary Outcome: Part 1: Renal Clearance (CLr) of TAK-117
Time Frame: Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Part-1: TAK-117 900 mg Capsules (9*100 mg Capsules) | Part-1: TAK-117 900 mg Tablets (3*300 mg Tablets)
Number analyzed (Participants) | 17 | 17
liter per hour (L/hr) | 0.314 (0.1179) | 0.311 (0.1304)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days (Day 46) after the last dose of study drug
Description: At each visit, investigator had to document any occurrence of adverse events and abnormal laboratory findings.Any event spontaneously reported by participant/observed by investigator was recorded,irrespective of relation to study treatment.Number at risk included those participants who have actually received the mentioned intervention during study.
Groups:
- Part-1: TAK-117 900 mg Capsules: TAK-117 9*100 mg, capsules (CTM), orally, once on Day 1 or 15 of intervention period.
- Part-1: TAK-117 900 mg Tablets: TAK-117 3*300 mg, tablets (NTM), orally, once on Day 1 or 15 of intervention period.
- Part-2: TAK-117 600 mg Fasted: TAK-117 2*300 mg, tablets (NTM), orally, once in a fasted state on Day 1 or 15 of intervention period.
- Part-2: TAK-117 600 mg Fed: TAK-117 2*300 mg, tablets (NTM), orally, with a standard high-fat breakfast, once on Day 1 or 15 of intervention period.
- Part-3: TAK-117 900 mg: TAK-117 3*300 mg, tablets (NTM), orally, once on Day 1.
- Part-3: Lansoprazole 30 mg: Lansoprazole 30 mg, capsule, orally, once daily from Day 10 to Day 14.
- Part 3: Lansoprazole 30 mg + TAK-117 900 mg: Lansoprazole 30 mg, capsule, orally, once daily on Day 15 along with TAK-117 3*300 mg, tablets (NTM), orally, once on Day 15.
Arm/Group | Part-1: TAK-117 900 mg Capsules | Part-1: TAK-117 900 mg Tablets | Part-2: TAK-117 600 mg Fasted | Part-2: TAK-117 600 mg Fed | Part-3: TAK-117 900 mg | Part-3: Lansoprazole 30 mg | Part 3: Lansoprazole 30 mg + TAK-117 900 mg
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/17 | 0/17 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/19 | 5/18 | 8/17 | 4/17 | 6/16 | 1/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part-1: TAK-117 900 mg Capsules (N=19) | Part-1: TAK-117 900 mg Tablets (N=18) | Part-2: TAK-117 600 mg Fasted (N=17) | Part-2: TAK-117 600 mg Fed (N=17) | Part-3: TAK-117 900 mg (N=16) | Part-3: Lansoprazole 30 mg (N=16) | Part 3: Lansoprazole 30 mg + TAK-117 900 mg (N=16)
Nausea (Gastrointestinal disorders) | 3 | 3 | 7 | 4 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.